CLINICAL TRIAL: NCT06336317
Title: Effect of infLuenza vaccInation After Myocardial INfArction on Cardiac inflammaTory responsE - a Randomized, Double-blind, Placebo-controlled, Trial (ELIMINATE Trial)
Brief Title: Effect of infLuenza vaccInation After Myocardial INfArction on Cardiac inflammaTory responsE
Acronym: ELIMINATE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: The Swedish Heart and Lung Association (Other); Örebro University, Sweden (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELIMINATE-2024
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Acute Myocardial Infarction; Cardiovascular Diseases; Inflammatory Response
Keywords: Coronary computed tomography angiography; Percutaneous coronary intervention; Influenza vaccine; Non ST-segment elevation myocardial infarction
MeSH Terms: conditions — Cardiovascular Diseases; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccination arm (Active Comparator): Influenza vaccine (Vaxigrip Tetra Sanofi Pasteur Europe).
  Interventions: Biological: Influenza vaccine
- Placebo arm (Placebo Comparator): Sodium Chloride (Placebo) Solution for infusion, 9mg/ml ATC code: B05BB01
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Influenza vaccine — VaxigripTetra Suspension for injection, 0,5ml prefilled syringe ATC code: J07BB02
  Arms: Vaccination arm
Biological: Placebo — Sodium Chloride Solution for infusion, 9mg/ml ATC code: B05BB01
  Arms: Placebo arm

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to investigate the immunological effects of influenza vaccination outside of the influenza season on arterial inflammation in patients with a recent acute myocardial infarction (AMI). The primary objective is to compare the effects of influenza vaccination to those of a placebo in reducing post-myocardial infarction coronary inflammation as measured by coronary computed tomography angiography (CCTA). The main questions it aims to answer are:

Does influenza vaccination reduce arterial inflammation as measured by CCTA at week 8 after percutaneous coronary intervention (PCI) in comparison to baseline? Does influenza vaccination modulate systemic inflammation as measured by blood biomarkers and in-vitro challenge tests at week 8 after PCI in comparison to baseline? Researchers will compare the effects of influenza vaccination with those of a placebo.

DETAILED DESCRIPTION:
Following informed consent patients are randomized in a 1:1 fashion to influenza vaccination or placebo up to 7 days following PCI. Blood tests for immune cell phenotyping and transcriptomic and proteomic analyses will be collected at baseline and 8 weeks after study inclusion. Patients will undergo CTCA at baseline (≤ 7 days of an AMI) and 8 weeks after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of non-ST-segment elevation myocardial infarction
* A finalized coronary PCI
* Male or non-fertile female subjects ≥18 years. (Females without childbearing potential, postmenopausal women and women with a history of hysterectomy or other medical conditions that preclude pregnancy)
* Written informed consent
* A CCTA can be scheduled within 7 days after PCI

Exclusion Criteria:

* Has received influenza vaccination within 6 months
* Other vaccination planned within 8 weeks (including covid-19 booster doses)
* Severe allergy to eggs or previous allergic reaction to influenza vaccine
* Cardiac surgery or staged PCI planned within 8 weeks
* Coronary stent involving the proximal RCA
* Suspicion of febrile illness or acute, ongoing infection
* Hypersensitivity to the active substances or ingredients of Vaxigrip or against any residues, such as eggs (ovalbumin or chicken proteins), neomycin, formaldehyde and octoxinol
* Subjects with endogenic or iatrogenic immunosuppression that may result in reduced immunization response
* Inability to provide informed consent
* Previous randomization in the ELIMINATE trial
* Any non-cardiovascular condition, e.g. malignancy, with a life expectancy of less than 1 year based on the investigator´s clinical judgement.
* Contraindication to coronary CT angiography (e.g., inability to lie flat, contraindication to glyceryl trinitrate, previous contrast allergy or contrast-induced nephropathy, severe renal impairment [eGFR <30 mL/min/1.73 m2])
* Atrial fibrillation
* Uncontrolled chronic inflammatory disease
* Unable to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The right coronary artery | Between baseline and 8 weeks follow up.
  Primary endpoint definition is a difference in pericoronary adipose tissue density (perivascular fat attenuation index) around the right coronary artery (RCA) measured by repeated CCTA imaging

SECONDARY OUTCOMES:
The whole coronary tree | Between baseline and 8 weeks follow up.
  Change from baseline in the average pericoronary adipose tissue density of the whole coronary tree (main epicardial arteries ≥2mm).
Ascending aorta | Between baseline and 8 weeks follow up.
  Change from baseline in the perivascular adipose tissue density of the ascending aorta
Interleukin 1 beta (IL-1β) | Between baseline and 8 weeks follow up.
  Difference in peripheral blood IL-1β concentrations
Tumor necrosis factor alpha (TNF-α) | Between baseline and 8 weeks follow up.
  Difference in peripheral blood TNF-α concentrations
Interleukin-2 receptor (IL-2r) | Between baseline and 8 weeks follow up.
  Difference in peripheral blood IL-2r concentrations
Interleukin Interleukin-6 (IL-6 ) | Between baseline and 8 weeks follow up.
  Difference in peripheral blood IL-6 concentrations
Ferritin | Between baseline and 8 weeks follow up.
  Difference in peripheral blood ferritin concentrations
Troponin-I | At 8 weeks follow up.
  Differences in peripheral blood troponin-I concentrations between study groups
N-terminal pro-B-type natriuretic peptide | At 8 weeks follow up.
  Differences in peripheral blood N-terminal pro-B-type natriuretic peptide concentrations between study groups

OTHER OUTCOMES:
Explorative endpoints | 8 weeks follow up
  Differences in peripheral blood immune cell signatures measured by mass cytometry (CyTOF), and proteomics (O-link) will be assessed in a subset of patients with and without reduction in coronary inflammation, measured by perivascular adipose tissue density on CCTA . Single cell RNA sequencing (sRNAseq) and measurements of cytokine profiles after in-vitro stimulation of peripheral blood mononuclear cells (PBMCs) will be performed in a subgroup of patients
Explorative endpoints | Baseline
  Exploratory proteomics by (O-link) from day 0 sampling will be performed in the whole study population to identify early biomarkers for prediction of residual inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Cajander, MD, Principal Investigator — Region Örebro län; Ole Frøbert, professor, Study Chair — Region Örebro län
Locations (1):
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No